CLINICAL TRIAL: NCT03281317
Title: Le Syndrome vasoplégique en Post-opératoire de Chirurgie Cardiaque: étude de Construction et de Validation d'un Score prédictif (Etude ISYVACC).
Brief Title: Vasoplegic Syndrome in Cardiac Surgery
Acronym: ISYVACC
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0014
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Vasoplegic Syndrome of Cardiac Surgery
Keywords: vasoplegicsyndrome; cardiac surgery; predictive risk score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vasoplasmic syndrome in cardiac surgery is one of the major postoperative complications.This syndrome is characterized by persistent low blood pressure despite an optimization of preload and inotropism.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery with extracorporeal circulation
* Patients covered by a social insurance system.
* Patients who have given oral consent to participate after full information

Exclusion Criteria:

* Cardiac graft.
* Preoperative ECMO / ECLS.
* Cardiac assistance.
* Minor,
* Patient deprived of liberty, or under safeguard of justice.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive cardiac surgical patients who meeet inclusion criteria with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 1113 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Vasoplegic syndrome | 30 days
  Patients suffering of vasoplegic syndrom defined by persitent arterial hypotension (MAP below70 mmHg) despite fluid rescucitation, normal or high cardiac output, and treated more than 4 hours with norepinephrine

SECONDARY OUTCOMES:
Post operative organ failure | 30 days
  every post opertaive organ failure: brain, digestive, renal, cardiac...
Arrythmia | 30 days
  atrial fibrillation, ventricular tachycardia, ventricular flutter
Inotropic use | 30 days
  dobutamine, levosimendan, phosphodiesterase
cardiac damage | 1 day
  troponine I release
Post operative Sepsis | 30 days
  postoperative sepsis: pneumonae, blood stream, mediastinis, urinary track, other
Hemorrhage | 30 days
  postopertaive blood loss defined by the Universal definition of perioperative bleeding
Blood transfusion | 30 days
  red blood cell transfusion, plaquette, plasma
ICU stays | 30 days
  Stay at ICU until patient discharge
Hospital stays | 30 days
  hospital stays until patient discharge
Death | one year
  Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Grégoire guinot.pierregregoire@chu-amiens.fr, Doctor, Study Director — guinot.pierregregoire@chu-amiens.fr; Paul Michel MERTES, Professor, Principal Investigator — CHU STRASBOURG; Jean-Luc Simon Jean-Baptiste FELLAHI, Professor, Principal Investigator — Hospices Civils de Lyon; FISCHER Marc Olivier, Professor, Principal Investigator — University Hospital, Caen; GIRARD Claude, Professor, Principal Investigator — CHU DIJON; Longrois Dan, Doctor, Principal Investigator — APHP, Paris; BESNIE Emmanuel, Doctor, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU Amiens Picardie, Amiens, France